CLINICAL TRIAL: NCT04381702
Title: Outcome After Laparoscopic Versus Open Pancreaticoduodenectomy: a Single Surgeon Experience
Brief Title: Outcome After Laparoscopic Versus Open Pancreaticoduodenectomy
Acronym: PaMIvOP
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0253
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Pancreatoduodenectomy
Keywords: Pancreatoduodenectomy; Benign or malign pathology; Mini-invasive approach; Morbimortality; Laparoscopic approach
MeSH Terms: interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with an open approach: Patients requiring pancreatoduodenectomy and operated with an open approach : All consecutive patients requiring pancreato-duodenectomies for benign or malignant pathology before the first laparoscopic pancreaticoduodenectomy.
  Interventions: Procedure: Pancreatoduodenectomy
- Patients with a laparoscopic approach: Patients requiring pancreatoduodenectomy and operated with a laparoscopic approach : All consecutive patients requiring pancreato-duodenectomies for benign or malignant pathology operated with a laparoscopic approach.
  Interventions: Procedure: Pancreatoduodenectomy

INTERVENTIONS:
Procedure: Pancreatoduodenectomy — Open or laparoscopic pancreato-duodenectomy with pancreatojejunal anastomosis

SUMMARY:
Aim of the study :

To determine the morbimortality of Laparoscopic pancreaticoduodenectomy (LPD) compared to the gold standard Open pancreaticoduodenectomy approach (OPD).

Methods :

This is a monocentric retrospective study based on a prospectively maintained clinical database. The study included 28 consecutive patients operated, between January 2016 and March 2019, of Laparoscopic pancreaticoduodenectomy (LPD) that we compared to 62 patients operated with the classical open approach by the same surgeon before the first laparoscopic resection at our institution.

DETAILED DESCRIPTION:
The progress achieved over the last 20 years and the growing experience of visceral surgeons in minimally invasive surgery allow us today to embark on increasingly complex surgeries.

Laparoscopic surgery has even become the gold standard approach for many interventions, whether for bariatric functional surgery, reflux surgery, pelvic static disorder surgery, but also for tumor surgery such as colorectal cancer, esophageal or tail of the pancreas.

However, there are still interventions which, due to their technical difficulty, do not find unanimous consensus among the international scientific community for a possible minimally invasive approach.

The close contact of the pancreatic gland with the splenomesaraic trunk making laparoscopic dissection difficult with risk of uncontrollable bleeding.

It seems, however, that the finesse of the dissection and coagulation instruments and the precision of today's optics make it possible to approach the head of the pancreas in completely satisfactory conditions.

Several centers around the world have developed the LPD technique with encouraging results in terms of perioperative mortality without showing any advantage over laparotomy.

At the Montpellier University Hospital we started performing Laparoscopic pancreaticoduodenectomy (LPD) at the beginning of 2016.

The aim of this study is to assess, on the one hand, the morbimortality and the quality of surgery linked to the development of this relatively new technique in a reference center for pancreatic surgery and on the other hand to assess a possible learning curve effect within our experience.

ELIGIBILITY:
Inclusion criteria:

- Pancreatoduodenectomy with pancreatojejunal anastomosis whatever the indication

Exclusion criteria:

-reject the study protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had Pancreatoduodenectomy with pancreatojejunal anastomosis whatever the indication
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Morbimortality of Laparoscopic pancreaticoduodenectomy (LPD) | 90 postoperative days
  Morbimortality of Laparoscopic pancreaticoduodenectomy (LPD) compared to the gold standard Open pancreaticoduodenectomy approach (OPD) :Overall morbidity (according to Clavien Dindo Classification)

SECONDARY OUTCOMES:
Number of lymph nodes removed | 14 postoperative days
  Number of lymph nodes removed
Margins of excision | 14 postoperative days
  Margins of excision R0, R1, R2

CONTACTS AND LOCATIONS:
Overall Officials: REGIS SOUCHE, Study Director — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided
NC